CLINICAL TRIAL: NCT07261566
Title: Assessment of Core Muscles Endurance, Lumber Curvature and Function in Smartphone-addicts With Chronic Nonspecific Low Back Pain
Brief Title: Assessment of Core Muscles Endurance, Lumber Curvature and Function in Smartphone-addicts With Nonspecific Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahd Ramadan, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/006095
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smartphone-addicted participants with chronic nonspecific low back pain.: This group included 33 smartphone-addicted participants with chronic nonspecific low back pain.
  Interventions: Other: non
- Smartphone-addicted participants without chronic nonspecific low back pain.: This group included 32 smartphone-addicted participants without chronic nonspecific low back pain.
  Interventions: Other: non

INTERVENTIONS:
Other:
Other: non

SUMMARY:
This study will attempt to assess the relation between, core muscle endurance, lumber spine curvature and function among smartphone-addicts university students with chronic nonspecific low back pain.

DETAILED DESCRIPTION:
It has been demonstrated that using a smartphone increases lumbar and cervical flexion. Moreover, using a smartphone while slouched increased the strain on the lumbar spine's muscles and capsular structures. Similarly, in other research, individuals with or without low back pain (LBP) experienced greater thoracic kyphosis and lumber lordosis following a brief period of smart phone use while seated.

In adults, mechanical LBP is frequently reported. Notably, there are several risk factors, including the excessive use of electronic and handheld electronic devices. Additionally, Back pain is linked to morphological changes in multifidus and erector spinae as a cross-sectional region.

In addition, core muscles are crucial for carrying out different motions or sustaining postures in day-to-day activities, particularly when sitting in a chair. They not only help to maintain endurance but also give the trunk muscles stability. Furthermore, weakness of the trunk muscles has been identified as a risk factor for LBP. Similarly, weak trunk muscular strength was linked to poor balance and functional performance. As a result, core muscle dysfunction leads to decreased trunk muscular strength, dynamic balance, and functional mobility.

Given these concerns, it is necessary to conduct further studies on the musculoskeletal problems linked to smartphone use. Therefore, all individuals experiencing musculoskeletal discomfort especially mechanical LBP should have their smartphone addiction level examined. Special attention should be given to addressing smartphone addiction and its musculoskeletal consequences on undergraduate students. Since young adults are a population that uses mobile phones often, they are an urgent group to investigate. However, no study has investigated the impact of smartphone use on the spinal and pelvic posture during standing and walking.

ELIGIBILITY:
Inclusion Criteria:

* University students who have been experiencing chronic nonspecific low back pain for a period of at least six months
* Both genders
* Smartphone addicted cut-off points for smartphone addiction at 31 for men and 33 for women in smartphone addiction scale short version
* Age is ranged from 18-25 years old

Exclusion Criteria:

* Patients will be excluded if they don't fulfil the inclusion criteria or if they have one of the following:
* Athletes
* Any history of spinal trauma or dysfunction
* Systemic disease presenting in the back (such as ankylosing spondylitis)
* Spinal deformity
* Leg length discrepancy
* History of spinal, abdominal or orthopedic surgery
* Patients who are under treatment with nonsteroidal anti-inflammatory drugs

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was conducted with a total of 65 participants. They were assigned into two groups, consisting of both genders with smartphone addiction according to the Smartphone Addiction Scale (SAS), and university students who had been experiencing chronic nonspecific low back pain for a period of at least six months
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Assessment of smartphone addiction | 8 weeks
  Smartphone addiction is examined using the Smartphone Addiction scale (SAS), which is a self-diagnosis instrument that identifies smartphone addicts. The final version included 33 items that revealed the presence of six subscales, including daily life disruption, positive anticipation, withdrawal, cyberspace-oriented connection, overuse, and tolerance.
  The items are assessed on a six-point Likert scale as follows: strongly disagree (1), disagree (2), weakly disagree (3), weakly agree (4), agree (5), and strongly agree (6). The total of the six subscales equals the SAS score, which ranges from 33 to 198; higher scores indicate more addicted behavior with smartphone use.
Assessment of lumbar spinal curvature | 8 weeks
  Kinovea software will be used to measure lumbar spinal curvature. The subject should be positioned in a sidelong stance without footwear, aligned with their back against a calibration plane, and their shoulders and elbows flexed at an angle of 90 degrees. Clearly delineate both earlobes on the subject Ascertain the critical reference points along the lumbar spine at 12 thoracic vertebra, third lumbar vertebra and first sacral vertebra. To ascertain the lordosis angle, identify the point on the lumbar spine that is nearest to the plumb line. Construct two lines that run parallel to the curvature of the lumbar region at both the superior and inferior aspects. Employ Kinovea to measure the angle formed at the intersection of these two lines. Deduct this measurement from 180° to derive the lordosis angle
Assessment of trunk anterior flexor test | 8 weeks
  During the trunk anterior flexor test, individuals sit with their hands over their chest, trunk flexed to sixty degrees, and knee flexed to ninety degrees, time starts when participants adopt the measured posture and ends when the trunk deviates from the 60º angle. The investigator uses the commands 'start' and 'stop' to begin and end the test, while an assisting investigator uses a stopwatch to record the times
Assessment of lateral musculature plank test | 8 weeks
  It will be applied for both sides. In the left lateral musculature plank test, participants' feet are placed one on top of the other, the right arm perpendicular to the floor, elbow lying on the mat, left arm across the chest, and left hand on the right shoulder. A similar position is used for the right lateral musculature plank test, with the left arm perpendicular to the floor. The investigator uses the commands 'start' and 'stop' to begin and end the test, while an assisting investigator uses a stopwatch to record the times. When the investigator observes an error in the line between the participants' trunk or lower body parts (thigh or shank), then time will be stopped.
Trunk posterior extensor test | 8 weeks
  Participants lie prone on an examination table for the trunk posterior extensor test, with both anterior superior iliac spines (ASISs) on the table's edge and their hands on the seat of a chair positioned in front of them. Assistance held the lower extremities above and below the participants' knees to secure the lower body. Time begins when participants establish a horizontal posture of the trunk, detach their hands from the chair and then cross them over their chest, and time will be stopped when participants are unable to maintain that position.
Assessment of back functional disability | 8 weeks
  The Oswestry Disability Index (ODI) is regarded as the 'gold standard' of low back functional outcome instruments. The questionnaire measures the level of impairment in ten activities of daily living: Pain intensity, Personal care, Lifting, Walking, Sitting, Standing, Sleeping, Sex (if applicable), Social, Travel. Each item has six statements that are evaluated from 0 to 5. The overall score is determined as a percentage, with 0% representing no disability and 100% indicating the highest level of disability

CONTACTS AND LOCATIONS:
Overall Officials: Rabab M Monged, PHD, Study Director — 6 October university; Salwa F Abdelmaged, Professor, Study Chair — Cairo University
Locations (1):
- Ahd Ramadan Mohamed, Giza, Egypt